CLINICAL TRIAL: NCT02884856
Title: Influence of Gender on Visual Shade Matching in Dentistry
Brief Title: Color Perception in Dentistry (CPD)
Acronym: CPD
Status: Completed | Type: Observational
Sponsor: Universidade de Passo Fundo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Ministerio de Economía y Competitividad, Spain (Other Government); Universidad de Granada (Other)
Responsible Party: Principal Investigator, Alvaro Della Bona, Senior Professor and Researcher, Universidade de Passo Fundo
Other Study IDs: 34553314.0.0000.5342
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Gender
Keywords: color; dentistry; gender
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Females observers (F): those with female gender characteristics
- Male observers (M): those with male gender characteristics

SUMMARY:
Visual shade matching (VSM) is the most common procedure to select an adequate shade in dentistry. This clinical procedure requires the use of a shade guide, being Vita Classical (VC) the most popular among the available guides. VSM is a subjective and inconsistent process with many observer related variables (e.g. color deficiency, experience, gender and eye fatigue) that can influence on the final color appearance. The gender influence on the accuracy of VSM is controversial.

The purpose of this study is to evaluate the VSM performed by female (F) and male (M) students, using VC shade guide, testing the null hypothesis that VSM is not influenced by gender.

DETAILED DESCRIPTION:
* Female and male observers will be analyzed.
* Human upper central incisors (UCI) will be shade matched to shade tabs from Vita Classical (VC) shade guide.
* The spectral reflectances from the four UCI and from the 16 VC shade tabs will be measured using a spectroradiometer (SP).
* Measurements will be performed over a gray background, inside a viewing booth and under D65 illuminant (diffuse/0º geometry).
* CIELAB coordinates (L*, a* and b*) will be calculated according to CIE D65 illuminant and CIE 2º Standard Observer.
* Two color difference metrics (CIELAB and CIEDE2000(2:1:1)) will be used to find the best option for each UCI, using VC shade guide.
* Data will be analyzed using descriptive statistics and McNemar test (α=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Dental students (DS) from University of Passo Fundo.
* DS with some knowledge and clinical experience with shade matching.
* DS from 20 to 35 years old.

Exclusion Criteria:

* DS with abnormal color vision.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Dental students from University of Passo Fundo (Brazil) and with some knowledge and clinical experience with shade matching will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Gender effect on visual shade matching | The study last for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Della Bona, Ph.D., Study Director — Universidade de Passo Fundo; Oscar E. Pecho, Ph.D., Principal Investigator — Universidade de Passo Fundo
Locations (1):
- Universidade de Passo Fundo, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abramov I, Gordon J, Feldman O, Chavarga A. Sex and vision II: color appearance of monochromatic lights. Biol Sex Differ. 2012 Sep 4;3(1):21. doi: 10.1186/2042-6410-3-21. PMID 22943488
- [Background] Capa N, Malkondu O, Kazazoglu E, Calikkocaoglu S. Evaluating factors that affect the shade-matching ability of dentists, dental staff members and laypeople. J Am Dent Assoc. 2010 Jan;141(1):71-6. doi: 10.14219/jada.archive.2010.0023. PMID 20045824
- [Background] Deeb SS. The molecular basis of variation in human color vision. Clin Genet. 2005 May;67(5):369-77. doi: 10.1111/j.1399-0004.2004.00343.x. PMID 15811001
- [Background] Della Bona A, Barrett AA, Rosa V, Pinzetta C. Visual and instrumental agreement in dental shade selection: three distinct observer populations and shade matching protocols. Dent Mater. 2009 Feb;25(2):276-81. doi: 10.1016/j.dental.2008.09.006. Epub 2008 Nov 18. PMID 19019420
- [Background] Donahue JL, Goodkind RJ, Schwabacher WB, Aeppli DP. Shade color discrimination by men and women. J Prosthet Dent. 1991 May;65(5):699-703. doi: 10.1016/0022-3913(91)90209-f. PMID 2051396
- [Background] Haddad HJ, Jakstat HA, Arnetzl G, Borbely J, Vichi A, Dumfahrt H, Renault P, Corcodel N, Pohlen B, Marada G, de Parga JA, Reshad M, Klinke TU, Hannak WB, Paravina RD. Does gender and experience influence shade matching quality? J Dent. 2009;37 Suppl 1:e40-4. doi: 10.1016/j.jdent.2009.05.012. Epub 2009 May 22. PMID 19520478
- [Background] Hugo B, Witzel T, Klaiber B. Comparison of in vivo visual and computer-aided tooth shade determination. Clin Oral Investig. 2005 Dec;9(4):244-50. doi: 10.1007/s00784-005-0014-3. Epub 2005 Oct 8. PMID 16215749
- [Background] Milagres V, Teixeira ML, Miranda ME, Osorio Silva CH, Ribeiro Pinto JR. Effect of gender, experience, and value on color perception. Oper Dent. 2012 May-Jun;37(3):228-33. doi: 10.2341/10-057-C. Epub 2012 Feb 15. PMID 22335300
- [Background] Paul S, Peter A, Pietrobon N, Hammerle CH. Visual and spectrophotometric shade analysis of human teeth. J Dent Res. 2002 Aug;81(8):578-82. doi: 10.1177/154405910208100815. PMID 12147751
- [Result] Pecho OE, Ghinea R, Alessandretti R, Perez MM, Della Bona A. Visual and instrumental shade matching using CIELAB and CIEDE2000 color difference formulas. Dent Mater. 2016 Jan;32(1):82-92. doi: 10.1016/j.dental.2015.10.015. Epub 2015 Nov 28. PMID 26631341